CLINICAL TRIAL: NCT05457062
Title: Study Based on Volatile Organic Compounds Analysis in Patients With Acute Upper Gastrointestinal Bleeding
Brief Title: Analysis the Vocs in Upper GI Bleeding Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: vocs in upper GI bleeding
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Upper GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — exhalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- large amount of bleeding: large amount of upper GI bleeding after EGD identified
- no bleeding: no upper GI bleeding after EGD identified
- small amount of bleeding: small amount of upper GI bleeding after EGD identified

SUMMARY:
This project aims to collect the exhaled breath of patients with acute upper gastrointestinal bleeding clinically, divide them into large, small and no bleeding groups according to the results of gastroscopy, analyze the characteristics of volatile organic compound components in exhaled breath, construct a discriminant model, and then analyze the sensitivity and specificity, and the target sensitivity and specificity reach more than 0.7, and formulate diagnostic criteria.

DETAILED DESCRIPTION:
Upper gastrointestinal bleeding is one of the most common gastrointestinal emergencies and has a high mortality rate. Its clinical manifestations are hematemesis and melena, gastroscopy is the gold standard for diagnosing upper gastrointestinal bleeding, but due to its expensive equipment, long training cycle of personnel, gastroscopy itself is an invasive operation, poor patient tolerance, high risk of examination, often lead to the diagnosis of upper gastrointestinal bleeding is not timely, missing the best treatment time. Volatile organic compound analysis in exhalation is based on the patient's metabolic component analysis technology, a new means of disease diagnosis, due to its advantages of convenient collection, non-invasive, rapid detection, etc., it has been applied in the diagnosis of various diseases such as drunken screening and Helicobacter pylori infection, but has not been studied in the diagnosis of upper gastrointestinal bleeding. This project aims to collect the exhaled breath of patients with acute upper gastrointestinal bleeding clinically, divide them into large, small and no bleeding groups according to the results of gastroscopy, analyze the characteristics of volatile organic compound components in exhaled breath, construct a discriminant model, and then analyze the sensitivity and specificity, and the target sensitivity and specificity reach more than 0.7, and formulate diagnostic criteria. This study will improve the timeliness of upper GI bleeding detection, which is of great significance for effectively reducing the mortality rate of upper GI bleeding.

ELIGIBILITY:
Inclusion Criteria: upper GI bleeding patients -

Exclusion Criteria: Severe cardiopulmonary disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: upper GI bleeding patients who will under go endoscopy examination
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
death in hospital | 6 weeks
  all cause death in hospital

SECONDARY OUTCOMES:
rebleeding | 5 days
  rebleeding in five days

CONTACTS AND LOCATIONS:
Locations (1):
- the Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China